CLINICAL TRIAL: NCT05190055
Title: Department of Neurosurgery, Chi-Mei Medical Center
Brief Title: Evaluation of Treatment Effect of Minimally Invasive Spinal Fusion Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chi Mei Medical Hospital (Other)
Responsible Party: Principal Investigator, Sher-Wei Lim, Director, Chi Mei Medical Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10508-J01
Record Dates: First submitted 2021-11-19; First posted 2022-01-13 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Spinal Fusion
Keywords: Spinal Fusion; Minimally invasive surgery

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimally invasive spinal fusion surgery (Experimental): A filler tube with an integrated threaded rod, which can be connected to a surgical drill, was used for rapid and continuous graft filling.
  Interventions: Device: bone graft delivery system/wiltrom interbody fusion system/wiltrom spinal fixation system
- traditional spinal fusion surgery (Active Comparator): Bone substitutes were filled in the disc space manually using a bone grafting funnel.
  Interventions: Device: wiltrom interbody fusion system/wiltrom spinal fixation system

INTERVENTIONS:
Device: bone graft delivery system/wiltrom interbody fusion system/wiltrom spinal fixation system — After receiving prophylactic antibiotics according to the local hospital protocol, the patients were generally anesthetized in a prone position. Paramedian or midline posterior sections were conducted, exposing the lumber vertebras encompassing the facet joints. The facet joints were removed, and decompression was performed. The diseased disc nucleus was then excised before filling in the bone substitutes. In the case of the device group, a novel filler tube with an integrated threaded rod, which can be connected to a surgical drill, A PEEK interbody fusion cage was then placed into the disc space followed by fixation with pedicle screws.
  Arms: Minimally invasive spinal fusion surgery
Device: wiltrom interbody fusion system/wiltrom spinal fixation system — After receiving prophylactic antibiotics according to the local hospital protocol, the patients were generally anesthetized in a prone position. Paramedian or midline posterior sections were conducted, exposing the lumber vertebras encompassing the facet joints. The facet joints were removed, and decompression was performed. The diseased disc nucleus was then excised before filling in the bone substitutes. For the control group, the bone substitutes were filled in the disc space manually using a bone grafting funnel. A PEEK interbody fusion cage was then placed into the disc space followed by fixation with pedicle screws.
  Arms: traditional spinal fusion surgery

SUMMARY:
Participants with lumbar spondylosis, degenerative disc disease, spondylolisthesis, scoliosis, or trauma undergoing elective Transforaminal lumbar interbody fusion (TLIF) were recruited. The follow-up period was 24 months for each participant. The eligible patients for this study should be above 18 years old with confirmed indication to TLIF through a posterior approach. Patients with an active infection, symptomatic osteoporosis, immature bone, pregnancy, active malignancy, and previous radiotherapy at the planned surgical site were excluded. Informed consent was signed by each participant before recruitment. We strictly followed the protocols of patient confidentiality and human subjects in the clinical trial implementation. The patients were blinded to the allocated surgical technique before the operation and during the follow-up period of two years. On the one hand, the doctor will assess the patient's physiological function recovery and imaging examinations (such as CT, MRI or X-ray) before and after the operation to understand the changes in the patient's pain index and the effect of intervertebral disc fusion after the operation; on the other hand, It also evaluates the quality of life and the degree of improvement of psychological emotions through the questionnaires of patients before and after surgery.

DETAILED DESCRIPTION:
After receiving prophylactic antibiotics according to the local hospital protocol, the patients were generally anesthetized in a prone position. Paramedian or midline posterior sections were conducted, exposing the lumber vertebras encompassing the facet joints. The facet joints were removed, and decompression was performed. The diseased disc nucleus was then excised before filling in the bone substitutes. For the control group, the bone substitutes were filled in the disc space manually using a bone grafting funnel. In the case of device group, a novel filler tube with integrated threaded rod, which can be connected to a surgical drill, was used for rapid and continuous graft filling (Figure 1). A polyethyletherketone (PEEK) interbody fusion cage was then placed into the disc space followed by fixation with pedicle screws. The treatment efficacy was assessed by clinical analysis based on the visual analogue scale (VAS) for radicular pain and the Oswestry Disability Index (ODI) questionnaire for low back pain. The VAS back and leg pain scores were measured preoperatively and postoperatively at 1, 3, 6, 12, and 24 months. The ODI questionnaires were taken preoperatively and postoperatively at 3, 6, 12, and 24 months. The bone graft delivery volume and the filling time during the surgery were measured to compare the efficiency of the two approaches.

The X-ray and computed tomography were performed prior to surgery and at 3-, 6-, 12-, and 24-monthspost-surgery for bone fusion assessment. The degree of bone fusion was classified into three grades. Grade I was defined as a complete fusion, union case, and grade II and III was defined as a partial union and a non-union case, respectively. Bone fusion volume was further determined by three-dimensional reconstruction images using ITK-SNAP software

ELIGIBILITY:
Inclusion Criteria:

spinal fusion procedures in skeletally mature patients with Degenerative Disc Disease (DDD) at one or two contiguous levels from L2 to S1. DDD is defined as discogenic back pain with degeneration of the disc confirmed by history and radiographic studies. These DDD patients may also have up to Grade I spondylolisthesis or retrolisthesis at the involved levels. Patients should have had six months of non-operative treatment prior to treatment with an intervertebral body fusion device.

Exclusion Criteria:

* Patients unsuitable for anesthesia
* Active systemic infection, infection or suspected latent infection localized to the site of the proposed implantation
* Excessive local inflammation
* Rapid joint disease, bone absorption, osteopenia
* Severe osteoporosis or osteopenia
* Morbid obesity
* Pregnancy
* Open wounds
* Patients have demonstrated allergy or foreign body sensitivity to any of the implant materials
* Any medical or surgical condition which would preclude the potential benefit of spinal implant surgery, surgery, such as the presence of tumors, congenital abnormalities, elevation of sedimentation rate unexplained by other diseases, elevation of white blood cell count (WBC), or marked left shift in the WBC differential count
* Patients whose activity, mental capacity, mental illness, alcoholism, drug abuse, occupation, or lifestyle may interfere with their ability to follow postoperative restrictions and who may place undue stresses on the implant during bony healing and may be at a higher risk of implant failure
* Any patient in which implant utilization would interfere with anatomical structures or expected physiological performance
* Any condition not described in the indications for use

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2015-03-25 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2023-02-26 (Estimated)

PRIMARY OUTCOMES:
Change of back pain at 24 months from baseline as measured by a 100 mm VAS scale | Preoperation and 24month post operation
  The back pain intensity on 100-mm VAS will be performed and recorded at Day 1 (within 48 hours before surgery as the Baseline) and 24th month.
Change of function at 24 months from baseline as measured by the 100 points Oswestry Disability Index (ODI) | Preoperation and 24month post operation
  The level of function on 100-point ODI will be performed and recorded at Day 1 (within 48 hours before surgery as the Baseline) and 24th month.

SECONDARY OUTCOMES:
Fusion Rates | 3, 6, 12, and 24 months
  Fusion rates for each product as evidenced by bridging bone via x-ray radiograph

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang KS, Chen CW, Yau RB, Liang HC, Ko CC, Kuo JR, Chio CC, Lim SW. A novel surgical technique in transforaminal lumbar interbody fusion by the bone graft delivery device: evaluation of therapeutic effect in patients with minimally invasive spine surgery. BMC Surg. 2022 Oct 26;22(1):366. doi: 10.1186/s12893-022-01773-y. PMID 36289500